CLINICAL TRIAL: NCT07146542
Title: Expression Pattern and Possible Clinical Significance of CD81 In Myeloid Leukemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Hesham Abdel Raheem, Assistant Lecturer, Assiut University
Other Study IDs: CD81 In Myeloid Leukemia
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Chronic Myeloid Leukemia
Keywords: CD81; AMl; CML; Myeloid; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients with myeloid leukemia

SUMMARY:
The goal of this study is to understand how the protein CD81 affects myeloid leukemia (especially AML) and whether it can help predict patient outcomes or guide treatment.

The main question it aims to answer:

Is high CD81 expression in myeloid leukemia cells linked to more aggressive disease, poorer treatment response, or shorter survival in patients?

Participants:

* Newly diagnosed myeloid leukemia patients (primary focus on AML)
* Bone marrow or blood samples will be collected during routine diagnostic procedures

DETAILED DESCRIPTION:
CD81, a cell surface protein belonging to the tetraspanin family, is overexpressed in 60-90% of acute myeloid leukemia (AML) patients and correlates with aggressive disease manifestations. Clinically, CD81-positive AML demonstrates elevated total leucocytic counts, increased lactate dehydrogenase (LDH) levels, higher bone marrow blast percentages, and a predominance in M1-M5 French-American-British (FAB) subtypes. Critically, this marker predicts adverse outcomes: reduced complete remission rates (12% vs. 24% in CD81-negative cohorts), higher relapse incidence (38% vs. 12%), and inferior overall, event-free, and relapse-free survival. Multivariate analyses confirm CD81 as an independent prognostic indicator, even within cytogenetically normal AML or NPM1-mutated subgroups.

Current AML risk stratification depends heavily on cytogenetic and molecular profiling (e.g., NPM1, FLT3-ITD). Nevertheless, 40-50% of patients lack identifiable high-risk genetic lesions, complicating clinical prognostication. Although flow cytometry enables rapid detection of CD81 surface expression, this biomarker remains underutilized in risk models despite its adverse impact mirroring established high-risk features. Mechanistically, CD81s involvement in metastasis and stem cell quiescence positions it as both a prognostic tool and a candidate therapeutic target.

Notably, CD81 expression remains uncharacterized in chronic myeloid leukemia (CML). Given CMLs distinct BCR::ABL1-driven pathogenesis and clinical trajectory from chronic phase to blast crisis, evaluating CD81s role may reveal novel biological insights or therapeutic vulnerabilities during disease progression.

ELIGIBILITY:
Inclusion Criteria:

* 1. Myeloid leukemia patients 2. Patients of both genders (Males and females) at any age 3. Cases are de novo (Not on treatment)

Exclusion Criteria:

* . Patients with other haematological neoplasms (ALL,CLL, plasma cell myeloma, etc)

  * Patients under any therapeutic intervention
  * Patients with current or previous other malignancies at time of diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Myeloid leukemia patients
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
expression of CD81 in patients with myeloid leukemia | baseline
  percentage of expression of CD81 in myeloid leukemia